CLINICAL TRIAL: NCT02102399
Title: Vocal Warm-up and Respiratory Training in Teachers: a Randomized Clinical Trial
Brief Title: Vocal Warm-up and Respiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Collaborators: Bahia State Secretariat of Education, Brazil (Unknown)
Responsible Party: Principal Investigator, Maria Lucia Vaz Masson, Maria Lucia Vaz Masson, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1152-9129
Record Dates: First submitted 2014-03-30; First posted 2014-04-02 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Voice Disorders
Keywords: Voice training; Education; Voice; Faculty
MeSH Terms: conditions — Voice Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vocal Warm-up (Experimental): Vocal Warm-up group performed 13 minutes of vocal warm-up exercises everyday before teaching over a course of 6 weeks, with one session exercise per day.
  Interventions: Behavioral: Vocal Warm-up
- Respiratory Muscle Training (Experimental): Respiratory Muscle Training group performed 13 minutes of Respiratory Muscle Training everyday before teaching over a course of 6 weeks, with one session exercise per day.
  Interventions: Behavioral: Respiratory Muscle Training

INTERVENTIONS:
Behavioral: Vocal Warm-up — Vocal Warm-up group performed 13 minutes of vocal warm-up exercises everyday before teaching over a course of 6 weeks, with one session exercise per day.
  Arms: Vocal Warm-up
Behavioral: Respiratory Muscle Training — Respiratory Muscle Training group performed 13 minutes of Respiratory Muscle Training everyday before teaching over a course of 6 weeks, with one session exercise per day.
  Arms: Respiratory Muscle Training

SUMMARY:
The purpose of this study is to verify the effects of two speech-pathology interventions: vocal warm-up and respiratory training in teachers who work in a public school of the city of Salvador-Bahia, with or without complaints of vocal disorders. It is a preventive study and the hypothesis is that both approaches can produce positive voice changes, but the Vocal Warm-up will produce the most significant changes.

DETAILED DESCRIPTION:
Randomized Clinical Trial where participants were allocated into groups: Vocal Warm-up (to perform exercises of resistance and flexibility for 13 minutes before teaching, during six weeks) and Respiratory Muscle Training (to perform exercises to strengthen the respiratory muscles through the use of incentive respiratory equipment. Five repetitions of exhales with an interval of thirty seconds between each one were performed. It was requested rest for two minutes, repeating the procedure four times with the total of five series. These exercises were performed for 13 minutes before teaching, during six weeks).

Outcomes analyzed: demographics and teaching activity characteristics; symptoms, habits and factors associated with voice disorders; self-reported voice handicap (Voice Handicap Index-VHI-10); vocal severity rating (Vocal Severity Scale); and acoustic parameters through the computerized acoustic voice analysis program VoxMetria (CTS Informatics).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60.
* No occurence of speech therapy simultaneously to the intervention

Exclusion Criteria:

* Professional voice use in another activity;
* Frequent use of alcohol and tobacco;
* Influenza and/or upper respiratory tract infections (eg, rhinitis, sinusitis, pharyngitis) during the period of participation in the research.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lucia V Masson, PhD, Principal Investigator — Federal University of Bahia; Lilian Paternostro, MS, Study Chair — Federal University of Bahia; Fernando M Carvalho, PhD, Study Director — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Pereira LP, Masson ML, Carvalho FM. Vocal warm-up and breathing training for teachers: randomized clinical trial. Rev Saude Publica. 2015;49:67. doi: 10.1590/S0034-8910.2015049005716. Epub 2015 Oct 9. PMID 26465664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The population sample was selected by convenience criteria. All the school's teachers were invited to participate and were selected according to eligibility criteria in the beginning of the study.
Groups:
- Vocal Warm-up: Vocal Warm up group performed 13 minutes of vocal warm-up exercises everyday before teaching over a course of 6 weeks, with one session exercise per day.
Period: Overall Study
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Started | 20 | 21
Completed | 14 | 17
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Population: Two different analyses were performed:
  1) Between-group (Vocal Warm-up vs. Respiratory Muscle Training) comparison analysis (n=31); 2a) Within-group (Respiratory Muscle Training Baseline vs Respiratory Muscle Post-test) comparison analysis (n=17); 2b) Within-group (Vocal Warm-up Baseline vs Vocal Warm-up Post-test) comparison analysis (n=14).
Groups:
- Vocal Warm-up: Vocal Warm up group was performed during 13 minutes of vocal warm-up exercises everyday before teaching over a course of 6 weeks, with one session exercise per day.
- Respiratory Muscle Training: Respiratory Muscle Training group was performed during 13 minutes of Respiratory Muscle Training everyday before teaching over a course of 6 weeks, with one session exercise per day.
- Total: Total of all reporting groups
Arm/Group | Vocal Warm-up | Respiratory Muscle Training | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (8.1) | 43.6 (11.4) | 44.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Voice Handicap Index (VHI-10)
Description: The voice handicap index (VHI) is a self-assessment questionnaire which quantifies the functional, physical and emotional impacts of a voice disorder on the quality of life. The VHI-10 is a reduced version and it consists of 10 questions about the severity of the voice problem perceived by the subject. It is presented as an ordinal scale (range 0-4) that indicates how frequently the subject has experienced the same situation (0 = never; 1 = almost never; 2 = sometimes; 3= almost always; 4 = always). Total VHI Score ranges from 0 (never) to 40 (always). Higher scores indicate greater voice handicap. Abnormal values > 11.
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Respiratory Muscle Training (Baseline); Respiratory Muscle Training (Posttest): Respiratory Muscle Training group performed 13 minutes of Respiratory Muscle Training everyday before teaching over a course of 6 weeks, with one session exercise per day.
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
units on a scale | 20.44 (13.70) | 13.82 (10.86)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.001, Wilcoxon's signed-rank test

2. Primary Outcome: Acoustic Analysis (Fundamental Frequency)
Description: The measurement of fundamental frequency directly reflects the rate of vibration of the vocal folds. The fundamental frequency term refers to the frequency of more occurrence of vocal fold vibration, featuring a certain production.
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Hertz (Hz)
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
Hertz (Hz) | 191.87 (43.35) | 185.71 (33.70)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.345, Wilcoxon's signed-rank test

3. Secondary Outcome: Post-treatment Questionnaire (Voice Symptoms Improvement)
Description: The post-treatment questionnaire was based on the original designed by Roy (2003) for assessing the teachers' perception of voice improvement and compliance with the intervention. Participants rated their extent of improvement on a 3-point Likert scale ("not at all/somewhat"; "moderate"; "a lot"). The questionnaire was applied only after the intervention. The answers were dichotomized in two categories ("moderate/a lot" and "not at all/somewhat"). The results were presented in frequency/percentage of subjects that answered "moderate/a lot" in each intervention.
Time Frame: After 6 weeks of intervention
Population: Between-group analysis
Measure: Number; unit: percentage of participants
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of participants | 64.3 | 11.8
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.003, Fisher Exact

4. Primary Outcome: Acoustic Analysis (Jitter)
Description: Jitter is the perturbation cycle-to-cycle of the fundamental frequency. High levels of jitter are normally associated with pathological voice. The instability of the fundamental frequency can be attributed to changes in size, shape or firmness of the vocal folds.
  Normal values must be < 0.6%.
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: percentage of jitter
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
percentage of jitter | 0.19 (0.14) | 0.45 (0.94)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.171, Wilcoxon's signed-rank test

5. Primary Outcome: Acoustic Analysis (Shimmer)
Description: The shimmer measures the amplitude's disturbance, e. g. how fast the amplitude changes on a sustained vowel for a few seconds. Shimmer high levels are normally associated with pathological voice. This can be attributed due to changes in size, shape or firmness of the vocal folds.
  Normal values < 6.5%.
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: percentage of shimmer
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
percentage of shimmer | 2.77 (0.94) | 4.19 (2.60)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.022, Wilcoxon's signed-rank test

6. Primary Outcome: Acoustic Analysis (Noise)
Description: Noise is the analysis of aperiodic components of the sound's signal. It is an important correlate of that the human ear considers voice disorders. Normal levels < 2.5 dB
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
Decibel (dB) | 0.72 (0.46) | 0.72 (0.44)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.451, Wilcoxon's signed-rank test

7. Primary Outcome: Acoustic Analysis (GNE)
Description: Glottal to Noise Excitation ratio (GNE) is an acoustic measurement to calculate the noise in a series of pulses produced by the oscillation of the vocal folds. This parameter is based on the hypothesis that resulting pulses of vocal fold collision generate a synchronous excitation of different frequency bands. Moreover, the noise produced by the vocal folds compressed generates uncorrelated excitations.
  Normal levels > 0.5 dB
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Respiratory Muscle Training (Baseline) | Respiratory Muscle Training (Posttest)
Number analyzed (Participants) | 17 | 17
Decibel (dB) | 0.88 (0.11) | 0.88 (0.11)
Statistical Analysis 1: Comparison: Respiratory Muscle Training (Baseline) vs Respiratory Muscle Training (Posttest); Test type: Superiority or Other; p = 0.477, Wilcoxon's signed-rank test

8. Primary Outcome: Voice Handicap Index (VHI-10) 2
Description: as for outcome 1
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vocal Warm-up (Baseline); Vocal Warm-up (Posttest): Vocal Warm-up group performed 13 minutes of vocal warm-up exercises everyday before teaching over a course of 6 weeks, with one session exercise per day.
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
units on a scale | 21.78 (17.44) | 13.04 (14.18)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.007, Wilcoxon's signed-rank test

9. Primary Outcome: Acoustic Analysis (Fundamental Frequency) 2
Description: as for outcome 2
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Hertz (Hz)
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
Hertz (Hz) | 196.21 (34.47) | 186.25 (31.53)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.049, Wilcoxon's signed-rank test

10. Primary Outcome: Acoustic Analysis (Jitter) 2
Description: as for outcome 4
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: percentage of jitter
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
percentage of jitter | 0.14 (0.11) | 0.10 (0.05)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.323, Wilcoxon's signed-rank test

11. Primary Outcome: Acoustic Analysis (Shimmer) 2
Description: as for outcome 5
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: percentage of shimmer
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
percentage of shimmer | 2.90 (0.85) | 3.10 (0.97)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.296, Wilcoxon's signed-rank test

12. Primary Outcome: Acoustic Analysis (Noise) 2
Description: as for outcome 6
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
Decibel (dB) | 0.69 (0.50) | 0.68 (0.50)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.776, Wilcoxon's signed-rank test

13. Primary Outcome: Acoustic Analysis (GNE) 2
Description: as for outcome 7
Time Frame: Baseline, 6 weeks
Population: Within-group analysis (pretest vs. posttest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Vocal Warm-up (Baseline) | Vocal Warm-up (Posttest)
Number analyzed (Participants) | 14 | 14
Decibel (dB) | 0.89 (0.12) | 0.92 (0.06)
Statistical Analysis 1: Comparison: Vocal Warm-up (Baseline) vs Vocal Warm-up (Posttest); Test type: Superiority or Other; p = 0.959, Wilcoxon's signed-rank test

14. Primary Outcome: Change in Voice Handicap Index (VHI-10)
Description: as for outcome 1
Time Frame: Baseline, 6 weeks
Population: Between-group analysis (mean difference posttest minus pretest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
units on a scale | -8.75 (10.13) | -6.61 (6.84)
Statistical Analysis 1: Comparison: Respiratory Muscle Training; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Change in Fundamental Frequency
Description: as for outcome 2
Time Frame: Baseline, 6 weeks
Population: Between-group analysis (mean difference posttest minus pretest)
Measure: Mean (Standard Deviation); unit: Hertz (Hz)
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
Hertz (Hz) | -9.96 (17.14) | -6.15 (26.11)
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)

16. Primary Outcome: Change in Jitter
Description: as for outcome 4
Time Frame: Baseline, 6 weeks
Population: Between-group analysis (mean difference posttest minus pretest)
Measure: Mean (Standard Deviation); unit: percentage of jitter
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of jitter | -0.02 (0.10) | 0.25 (0.89)
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

17. Primary Outcome: Change in Shimmer
Description: Shimmer measures the amplitude perturbations, e. g. how fast the amplitude changes on a sustained vowel for a few seconds. Shimmer high levels are normally associated with pathological voice. This can be attributed due to changes in size, shape or firmness of the vocal folds. Normal values < 6.5%
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of shimmer
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of shimmer | 0.20 (0.89) | 1.41 (2.30)
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)

18. Primary Outcome: Change in Noise
Description: as for outcome 6
Time Frame: Baseline, 6 weeks
Population: Between-group analysis (mean difference posttest minus pretest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
Decibel (dB) | -0.01 (0.14) | -0.004 (0.67)
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney)

19. Primary Outcome: Change in GNE
Description: as for outcome 7
Time Frame: Baseline, 6 weeks
Population: Between-group analysis (mean difference posttest minus pretest)
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
Decibel (dB) | 0.02 (0.13) | 0.001 (0.67)
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Post-treatment Questionnaire (Voice Clearer)
Description: as for outcome 3
Time Frame: After 6 weeks of intervention
Population: Between-group analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of subjects | 50 | 17.7
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.120, Fisher Exact

21. Secondary Outcome: Post-treatment Questionnaire (Easier to Talk)
Description: as for outcome 3
Time Frame: After 6 weeks of intervention
Population: Between-group analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of subjects | 57.2 | 17.7
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.030, Fisher Exact

22. Secondary Outcome: Post-treatment Questionnaire (Compliance With Intervention)
Description: The post-treatment questionnaire was based on the original designed by Roy (2003) for assessing the teachers' perception of voice improvement and compliance with the intervention. Participants rated their degree of compliance on a 3-point Likert scale ("not at all/somewhat"; "moderate"; "a lot"). The questionnaire was applied only after the intervention. The answers were dichotomized in two categories ("moderate/a lot" and "not at all/somewhat"). It was considered compliance the answers "moderate" and "a lot" in comparison of "not at all/somewhat", considered as no compliance. The results were presented in frequency/percentage of subjects in each intervention.
Time Frame: After 6 weeks of intervention
Population: Between-group analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Number analyzed (Participants) | 14 | 17
percentage of subjects | 100 | 76.5
Statistical Analysis 1: Comparison: Vocal Warm-up vs Respiratory Muscle Training; Test type: Superiority or Other; p = 0.107, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6-week intervention period
Description: The participants were monitored daily throughout the intervention period.
Arm/Group | Vocal Warm-up | Respiratory Muscle Training
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
Small and not probabilistic sample; type I error; type II error; strike in the last week of the study; healthy worker effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No